CLINICAL TRIAL: NCT06731686
Title: Single-center Retrospective Study : Developmental Trajectories of Children Born Prematurely Before 32 Weeks Assessed With the Revised Brunet Lézine Scale at 1, 2 and 3 Years
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Creteil (Other)
Responsible Party: Sponsor
Other Study IDs: PREMADEV
Record Dates: First submitted 2024-03-25; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Premature Birth
Keywords: Developmental trajectories; Revised Brunet Lézine; movement and posture; language; socialization; coordination
MeSH Terms: conditions — Premature Birth; Language | interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Retrospective study — Collection of children's datas

SUMMARY:
This study will assess professionals in the CHI Créteil neonatal department and the Val de Marne perinatal network to gain a better understanding of the developmental trajectories of children hospitalized at the CHI Créteil, with a view to optimizing their care in the long term

ELIGIBILITY:
Inclusion Criteria:

* Children born at CHI Créteil between 2012 and 2022, included in the Val de Marne perinatal network.
* Children seen in pediatrician-psychomotor consultation with assessment by the BLR scale at 1 year AC.

Exclusion Criteria:

* Children born with a term of birth ≥ 32 weeks + 1 day.
* Child removed from the Val de Marne perinatal network monitoring from the age of 1 year AC: Death or parental decision.
* Children presenting with cerebral palsy, blindness or deafness at the age of 1 year AC.

Ages: 2 Months to 32 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children born prematurely before 32 weeks
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-06-17 (Actual); Study Completion 2024-06-17 (Actual)

PRIMARY OUTCOMES:
Overall DQ obtained on the BLR scale at 1, 2 and 3 years, collected by the psychomotor therapists at CHI Créteil. | 1, 2 and 3 years

SECONDARY OUTCOMES:
Analysis of the 4 sub-scores (movement and posture, language, socialization, coordination) obtained on the BLR scale at 1, 2 and 3 years, collected by the psychomotor therapists at CHI Créteil. | 1,2 and 3 years
Analysis of family socio-demographic data : level of education | 1,2 and 3 years
Analysis of family socio-demographic data : age of parents | 1,2 and 3 years
Analysis of birth data : term | 1, 2 and 3 years
Analysis of birth data : weight | 1,2 and 3 years
Analysis of duration of hospitalization | 1,2 and 3 years
Evaluate the concordance of BLR scale at 5 years with the measurement scores (not validated) used by the Val de Marne perinatal network (and all the Ile de France perinatal networks) filed out during the same consultations | 5 years
Evaluate the concordance of BLR scale at 5 years with the measurement scores (not validated) used by the Val de Marne perinatal network (and all the Ile de France perinatal networks) filed out during the same consultations | 1,2 and 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- CHI Créteil, Créteil, France

IPD SHARING:
Plan to Share IPD: No